CLINICAL TRIAL: NCT02091765
Title: A Randomized Study of an Internet-based Cognitive Behavioral Therapy Program for Sexuality and Intimacy Problems in Women Treated for Breast Cancer.
Brief Title: RCT of an Internet-based CBT Program for Sexuality and Intimacy Problems in Women Treated for Breast Cancer
Acronym: KIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other); Pink Ribbon Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKI 2012-5388 / NL44153.031.13
Record Dates: First submitted 2014-03-07; First posted 2014-03-19 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2016-10

CONDITIONS: Sexual Dysfunction; Intimacy Problems; Breast Cancer Survivors
Keywords: Sexual dysfunction; Intimacy problems; Breast cancer survivors; Internet-based; Cognitive behavioral therapy
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimal intervention control group (No Intervention): Women who are assigned to the control group will be contacted by telephone by a member of the study staff to inform them about this allocation. They will receive a booklet per mail that addresses 80 questions about sexuality and cancer. Six weeks later, they will receive an empathetic phone call from one of the sexologists, during which there is also time available to discuss further questions the participants may have concerning sexuality and cancer. The purpose of keeping in contact with the control group, as opposed to a pure waiting list control group, is creating the opportunity to provide some control for a possible attention placebo-effect. The final questionnaire will be completed twenty weeks post study entry, after which women will be given the opportunity to undergo the internet-based cognitive behavioral program.
- Internet-based cognitive behavioral therapy (Experimental): Each woman who is allocated to the intervention group is assigned a personal sexologist (therapist) who guides her through the internet-based cognitive behavioral therapy (CBT) program and provides feedback on the homework assignments. The CBT program comprises a maximum of ten treatment modules that can be used in varying order. Each module contains three interventions and a personal evaluation form to report on the intervention. Each intervention comprises the following elements: 1) introduction, 2) psycho-education about symptoms, 3) "homework" assignments (e.g. relaxation techniques (pelvis); discuss intimacy with partner; sensate focus) and 4) reporting back to the therapist and receiving feedback on the "homework" assignments. Each week there are two "practice" sessions of 30 minutes each and one hour per week to report on/evaluate the intervention. The therapy has a mean duration of 20 weeks.
  Interventions: Behavioral: Internet-based cognitive behavioral therapy.

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioral therapy.
  Arms: Internet-based cognitive behavioral therapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and cost-effectiveness of an internet-based cognitive behavioural therapy program in alleviating problems with intimacy and sexuality in women treated for breast cancer.

DETAILED DESCRIPTION:
Background. Breast cancer is the most common cancer among women in the Netherlands, with an incidence of 71 per 100.000 person-years, and a lifetime risk of 10%. Currently, 85% of women with breast cancer live longer than 5 years, and 75% 10 years or longer(1,2). As a result, more interest and research has focused on the health-related quality of life (HRQL) of breast cancer survivors, including issues of sexuality and intimacy. Compelling evidence has established that sexual dysfunction is a prevalent, long term complication of breast cancer and its treatment (3,4-11). Overall, approximately 50% of breast cancer survivors report some form of sexual dysfunction as a result of treatment(6,10,13-15). Frequently reported problems regarding intimacy and sexuality include decreased sexual desire (23-64%), decreased arousal or lubrication (20-48%), anorgasmia (16-36%) and dyspareunia (35-38%)(10). Hill et al. report that over 40% of the breast cancer and gynaecological cancer survivors in their study expressed interest in receiving professional sexual health care(15). However, there is a significant discrepancy between the self-reported need for professional sexual health care and the actual uptake of care(16). Hill et al.(15) reported that, although over 40% of their sample expressed interest in receiving professional care, only 7% had ever actually sought such care. Although sexual functioning is an important issue, it may be difficult for women to initiate discussion with their general practitioner or medical specialist. Health care professionals may also be reluctant to query about sexual problems, due to time constraints, embarrassment, and/or lack of experience and communication skills in this area(16,17). Many women consider face-to-face sexual counselling to be confronting, and see internet-based interventions as a less threatening and more acceptable approach(18,19). There is growing evidence that internet-based cognitive behavioural therapy (CBT) can effectively treat a range of psychosocial problems, including anxiety, depression and PTSD(20,21). More recently, internet-based cognitive behavioural therapy programs for sexual dysfunction have been developed, typically paralleling the content of face-to-face therapy, with studies showing the efficacy of these internet-based programs in improving sexual functioning(22-25).

Design. This pragmatic clinical trial will employ a prospective, randomized design with one intervention group and a control group. Potentially eligible patients will be identified through the hospital registries. These patients will be sent a letter signed by their treating/former surgeon, together with an informational brochure about the study and possible cancer-related intimacy and sexuality problems. Women who are potentially interested in participating in the study will be asked to indicate this on the enclosed response card. Women who are not interested in participation will be requested to return the response card to indicate their motive(s) for not being able to participate. Women who are not interested in participation or who do not respond to the invitation to participate in the study will not be contacted again. If interested, women are asked to write down their contact information. Those women who return the questionnaire will be contacted by telephone by one of the members of the study staff to inform them more thoroughly about the study purpose and procedures. At this time, additional questions will be posed regarding current treatment of sexuality/intimacy problems, current participation in a research trial with a focus on alleviating sexuality/intimacy problems, access to internet, date of breast cancer diagnosis, and completion/continuation of the different parts of treatment of breast cancer (chemotherapy, radiation therapy, endocrine treatment).

Those women who remain interested in the study and who appear to be eligible will undergo an intake evaluation by telephone with a sexologist who will carry out a more extensive diagnostic interview in order to determine final eligibility of the woman for the internet-based cognitive behavioral therapy program. Questions will be asked about problems with sexuality and intimacy and relationship/marriage.

If the woman meets final eligibility criteria, she will receive a baseline questionnaire, together with an informed consent form. The questionnaire will assess sociodemographic and medical background variables, and the primary (sexuality and intimacy problems) and secondary study outcomes (body image, menopausal symptoms, marital functioning, psychological distress and health-related quality of life). In total, 160 consenting women will be randomized to either the intervention group (n = 80), or to a control group (n = 80) using the minimization technique, with primary surgery (breast conserving treatment; mastectomy without reconstructive surgery; mastectomy with reconstructive surgery), menopausal status (premenopausal; postmenopausal), current endocrine treatment for breast cancer (yes; no), and time since breast cancer diagnosis (<1 year; 1-3 yrs; 3-5 yrs) as stratification variables. Women allocated to the intervention group will be asked to complete a battery of questionnaires assessing primary and secondary outcomes at four points in time: ten weeks after the start of the CBT program (T1), and at post-treatment (T2; to achieve an equivalent average assessment time for both study groups, women in the intervention group complete T2 post-treatment, but always between 20 and 24 weeks after start of therapy. Women who finish the CBT prior to 20 weeks complete T2 20 weeks after start of therapy). The last two questionnaires are completed 3-months after completion of therapy (T3) and 6 months after T3 (T4). The control group is not asked to complete T3 or T4, but rather is given the opportunity to undergo the intervention following completion of T2. This was done because it was not deemed ethically acceptable to withhold the intervention from women in the control group for the prolonged period of time that would be required if they were to be first asked to complete all follow-up sessions (i.e., approximately one year after study enrollment). To minimize respondent burden, the T4 questionnaire only includes questionnaires assessing the primary outcome measures.

Control group. Women who are assigned to the control group will be contacted by telephone by a member of the study staff to inform them about this allocation. These women will receive a booklet per mail that addresses 80 questions about sexuality and cancer. Six weeks later, women in the control group will receive an empathetic phone call from one of the sexologists, during which there is also time available to discuss further questions the participants may have concerning sexuality and cancer. The purpose of keeping in contact with the control group, as opposed to a pure waiting list control group, is creating the opportunity to provide some control for a possible attention placebo-effect. Ten weeks post study entry, women in the control group will be asked to complete the first follow-up questionnaire. After completion of the questionnaire, women in the control group will be telephoned by a member of the study staff for another empathetic conversation. Women in the control group will complete a final questionnaire twenty weeks post study entry, after which they will be given the opportunity to undergo the internet-based cognitive behavioral program.

Intervention group. For women allocated to the intervention group, the sexologist will develop a tailored treatment plan, consisting of a maximum of 10 treatment modules (see below for a more detailed description of the intervention). The therapist has received specialized training in the nature of breast cancer and its treatment, in general, and more specifically sexuality and intimacy issues associated with breast cancer and its treatment. Each woman is assigned a personal sexologist (therapist) who guides her through the internet-based CBT program and provides feedback on the homework assignments. Contact with the therapist is fully web-based, via a secured website. The CBT program comprises a maximum of ten treatment modules that can be used in varying order. The choice of modules to be used by any given woman is based on the information obtained via the screening by telephone and the intake evaluation by the therapist. Each module contains three interventions and a personal evaluation form to report on the intervention. Each intervention comprises the following elements: 1) introduction, 2) psycho-education about symptoms, 3) "homework" assignments (e.g. relaxation techniques (pelvis); discuss intimacy with partner; sensate focus) and 4) reporting back to the therapist and receiving feedback on the "homework" assignments. Each week there are two "practice" sessions of 30 minutes each and one hour per week to report on/evaluate the intervention. The therapy has a mean duration of 20 weeks.The modules include: (1) "Put your problem into words" where the client describes her problems, is asked to distinguish between feelings, thoughts, and behaviors, and learns about what intimacy is and how it interplays with sexuality, the sexual response curve and the most common (psycho)sexual problems; (2) "How is my relationship doing?" in which the client explores how intimate the relationship actually is, becomes aware of the amount of quality time spent with the partner, receives psycho-education about sex and intimacy, the importance of open communication with the partner, and advice on how to improve open communication; (3) "Sex and my body" during which the client first experiences sensate focus therapy (targeted at becoming more comfortable with one's own body and achieving (non) sexual intimacy with one's partner physically and emotionally); (4) "Focus my attention" in which the client receives task concentration training to learn to focus her attention on sexual experiences; (5) "Explore my body" in which sensate focus therapy is further used, and the client writes about her experiences with the homework exercises within a cognitive behavioral framework (with particular focus on inhibiting thoughts); (6 & 7) "Discovering my sexual arousal feelings (versions for the woman and for her partner) in which psycho-education is provided about genital stimulation, sexual techniques, etc., and how to discuss sexual feelings with the partner; (8) "Change my thoughts" that involves cognitive restructuring to promote adaptive thoughts; (9) "My sexual preferences" in which the client talks about her sexual preferences with her partner, and makes an action plan for behavior change; and (10) "Relapse prevention" in which the client writes about her former automatic behavior and the risk factors for relapse, after which a plan of action is made in case of a relapse.

Study measures. The primary outcomes (sexuality and intimacy problems) are measured using the Sexual Activity Questionnaire, Female Sexual Functioning Scale, Female Sexual Distress Scale and the Personal Assessment of Intimacy in Relationships. Secondary outcomes measures include QLQ-BR23 (body image), FACT-ES (menopausal symptoms), Maudsley Marital Questionnaire (marital functioning), Hospital Anxiety and Depression Scale (psychological distress) and MOS SF-36 (health-related quality of life).

Program adherence. Women who do not complete their tailored internet-based therapy program will be asked to indicate the reason(s) for their discontinuation (e.g., illness, lack of motivation, burden, etc.). Every effort will be made to obtain a final, post-intervention assessment for all women, regardless of whether they do or do not complete their therapy. This will facilitate a maximum sample size for the primary, 'intention-to-treat' analysis of between-group differences over time. Additionally, all women, including those in the control group, will be asked if, during the period of the study, they pursued any (other) activities relating to their sexual and intimacy issues.

Patients' evaluation of the intervention program. At the end of their treatment, women in the intervention group will be asked about their experience with the module, the homework assignments, and the feedback received from the therapist. Additionally, immediate post-treatment, these women will be asked whether they would suggest any changes to the program, and if they would recommend it to other women experiencing similar problems.

Semi-structured interview. A subset of women (approximately 15 from the intervention group) will be asked to participate in a telephone interview. This semi-structured interview will cover the same topic areas as addressed by the self-report questionnaire, allowing women to provide feedback in a more narrative form about their sexual wellbeing and their experience with the CBT program. Women will also be asked if their partner would be willing to share his/her experience with the program (where applicable). The interview protocol has been developed and pilot-tested during the preparatory phase of the study.

Sample size and statistical power calculations. The prospective study design will allow for testing of the main effect of the internet-based intervention program. The SAQ, FSFI, FSFS and PAIR Inventory are the primary outcome measures on which sample size calculations are based. Specifically, the difference between the SAQ, FSFI and FSDS scores at baseline, mid-treatment (e.g. after 10 weeks), post-treatment (e.g. after 20 weeks), at 3 months follow-up (T3) and at 9 months follow-up (T4) will be calculated for each patient, and these changes will be the primary endpoints of the study. The mean of these differences in scores will be compared with the minimal intervention control group.

With a total sample of 130 women (65 per group), and under the assumption of no interaction, the study will have 80% power to detect an effect size of 0.5 for the main effects of the web based intervention program, with the p value set at 0.05.

160 women will be recruited into the study, to allow for an attrition rate of approximately 20% (i.e., women who discontinue participation in the study entirely, including failure to complete all follow-up questionnaires). Those women who discontinue participation in one of the groups but complete the follow-up assessments will be included in the intention-to-treat analysis.

Statistical analyses. Analysis will first be performed to evaluate the comparability of the intervention and control group at baseline in terms of sociodemographic and clinical characteristics. Student's t-test or appropriate non-parametric statistics will be used, depending on the level of measurement. If, despite the stratified randomization procedures, the groups are found not to be comparable on one or more background variables, those variables will be employed routinely as covariates in subsequent analyses.

Questionnaire scores will be calculated according to published scoring algorithms. Between-group differences over time in mean scores will be tested using multilevel analysis. Effect sizes will be calculated using standard statistical procedures. Effect sizes of 0.2 will be considered as small, 0.5 moderate, and 0.8 large. Effect sizes of approximately 0.4 will be considered as clinically relevant. All analysis will, to as great an extent as possible, be conducted on an intention-to-treat basis. The variables used in the minimization procedure will be employed as covariates. Per protocol analyses will also be carried out (as a secondary analysis), comparing women who meet minimal compliance levels (to be defined) with the program to the control group. We will also use correlation analyses to examine the relationship between degree of program adherence, partner involvement, and program effect. As indicated previously, the SAQ, FSFI, FSDS and PAIR inventory will be used as the primary study endpoints, and the remaining measures will be considered as secondary endpoints. For the analysis of these latter variables, appropriate statistical (p value) adjustments will be made for multiple testing. Since the sample size will not provide sufficient power to conduct subgroup analyses, an interaction term (group x time since diagnosis) will be added to the analyses. The semi-structured interview data will be transcribed and content analyzed to extract narrative, qualitative information about the women's sexual and intimacy problems and, where relevant, their experience with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Woman.
* Between 18 and 65 years of age.
* Diagnosis of histologically confirmed primary breast cancer.
* Received treatment in one of the participating hospitals.
* Completed treatment for breast cancer(with the exception of endocrine therapy).
* Diagnosis of breast cancer between 6 months and 5 years prior to study entry.
* Disease-free at time of study entry.
* Presence of sexuality and intimacy problems.

Exclusion Criteria:

* Lacks basic proficiency in Dutch.
* No access to the internet.
* Serious cognitive or psychiatric problems (i.e. depression, alcohol dependency, or psychotic disorders).
* Severe relationship problems for which the internet-based program is not designed (and which need to be addressed prior to undergoing sex therapy).
* Participation in a concurrent therapy program to alleviate sexuality/intimacy problems.
* Treated for another type of cancer beside breast cancer (with the exception of cervical carcinoma in situ and basal cell carcinoma).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-12; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Sexuality problems | Baseline
  Sexuality problems are assessed using the Sexual Activity Questionnaire, Female Sexual Function Scale, and Female Sexual Distress Scale.
Intimacy problems. | Baseline
  Intimacy problems are assessed using the Personal Assessment of Intimacy in Relationships (PAIR) Inventory.
Sexuality problems | T1: 10 weeks after start of therapy (intervention group) or 13 weeks after completion of baseline (control group)
  Sexuality problems are assessed using the Sexual Activity Questionnaire, Female Sexual Function Scale, and Female Sexual Distress Scale.
Sexuality problems | T2: 20-24 weeks after start of therapy (intervention group) or 23 weeks after completion of baseline (control group)
  Sexuality problems are assessed using the Sexual Activity Questionnaire, Female Sexual Function Scale, and Female Sexual Distress Scale.
Sexuality problems | T3: 3 months after T2 (intervention group)
  Sexuality problems are assessed using the Sexual Activity Questionnaire, Female Sexual Function Scale, and Female Sexual Distress Scale.
Intimacy problems. | T1: 10 weeks after start of therapy (intervention group) or 13 weeks after completion of baseline (control group)
  Intimacy problems are assessed using the Personal Assessment of Intimacy in Relationships (PAIR) Inventory.
Intimacy problems. | T2: 20-24 weeks after start of therapy (intervention group) or 23 weeks after completion of baseline (control group)
  Intimacy problems are assessed using the Personal Assessment of Intimacy in Relationships (PAIR) Inventory.
Intimacy problems. | T3: 3 months after T2 (intervention group)
  Intimacy problems are assessed using the Personal Assessment of Intimacy in Relationships (PAIR) Inventory.
Sexuality problems | T4: 6 months after T3 (intervention group)
  Sexuality problems are assessed using the Sexual Activity Questionnaire, Female Sexual Function Scale, and Female Sexual Distress Scale.
Intimacy problems | T4: 6 months after T3 (intervention group)
  Intimacy problems are assessed using the Personal Assessment of Intimacy in Relationships (PAIR) Inventory.

SECONDARY OUTCOMES:
Body image. | Baseline
  Body image is assessed using the QLQ-BR23.
Menopausal symptoms. | Baseline
  Menopausal symptoms are assessed using the FACT-ES.
Marital functioning. | Baseline
  Marital functioning is assessed using the Maudsley marital Questionnaire.
Psychological distress | Baseline
  Psychological distress is assessed using the Hospital Anxiety and Depression Scale.
Health-related quality of life | Baseline
  Health-related quality of life is assessed using the MOS SF-36.
Body image. | T1: 10 weeks after start of therapy (intervention group) or 13 weeks after completion of baseline (control group)
  Body image is assessed using the QLQ-BR23.
Body image. | T2: 20-24 weeks after start of therapy (intervention group) or 23 weeks after completion of baseline (control group)
  Body image is assessed using the QLQ-BR23.
Body image. | T3: 3 months after T2 (intervention group)
  Body image is assessed using the QLQ-BR23.
Menopausal symptoms. | T1: 10 weeks after start of therapy (intervention group) or 13 weeks after completion of baseline (control group)
  Menopausal symptoms are assessed using the FACT-ES.
Menopausal symptoms. | T2: 20-24 weeks after start of therapy (intervention group) or 23 weeks after completion of baseline (control group)
  Menopausal symptoms are assessed using the FACT-ES.
Menopausal symptoms. | T3: 3 months after T2 (intervention group)
  Menopausal symptoms are assessed using the FACT-ES.
Marital functioning. | T1: 10 weeks after start of therapy (intervention group) or 13 weeks after completion of baseline (control group)
  Marital functioning is assessed using the Maudsley Marital Questionnaire.
Marital functioning. | T2: 20-24 weeks after start of therapy (intervention group) or 23 weeks after completion of baseline (control group)
  Marital functioning is assessed using the Maudsley Marital Questionnaire.
Marital functioning. | T3: 3 months after T2 (intervention group)
  Marital functioning is assessed using the Maudsley Marital Questionnaire.
Psychological distress | T1: 10 weeks after start of therapy (intervention group) or 13 weeks after completion of baseline (control group)
  Psychological distress is assessed using the Hospital Anxiety and Depression Scale.
Psychological distress | T2: 20-24 weeks after start of therapy (intervention group) or 23 weeks after completion of baseline (control group)
  Psychological distress is assessed using the Hospital Anxiety and Depression Scale.
Psychological distress | T3: 3 months after T2 (intervention group)
  Psychological distress is assessed using the Hospital Anxiety and Depression Scale.
Health-related quality of life | T1: 10 weeks after start of therapy (intervention group) or 13 weeks after completion of baseline (control group)
  Health-related quality of life is assessed using the MOS SF-36.
Health-related quality of life | T2: 20-24 weeks after start of therapy (intervention group) or 23 weeks after completion of baseline (control group)
  Health-related quality of life is assessed using the MOS SF-36.
Health-related quality of life | T3: 3 months after T2 (intervention group)
  Health-related quality of life is assessed using the MOS SF-36.

CONTACTS AND LOCATIONS:
Overall Officials: Neil K. Aaronson, PhD, Principal Investigator — The Netherlands Cancer Institute; Jacques J. van Lankveld, PhD, Principal Investigator — Open University, the Netherlands; Hester S. Oldenburg, PhD, Principal Investigator — The Netherlands Cancer Institute; Daniela Hahn, MSc, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

REFERENCES:
- [Background] Coleman MP, Quaresma M, Berrino F, Lutz JM, De Angelis R, Capocaccia R, Baili P, Rachet B, Gatta G, Hakulinen T, Micheli A, Sant M, Weir HK, Elwood JM, Tsukuma H, Koifman S, E Silva GA, Francisci S, Santaquilani M, Verdecchia A, Storm HH, Young JL; CONCORD Working Group. Cancer survival in five continents: a worldwide population-based study (CONCORD). Lancet Oncol. 2008 Aug;9(8):730-56. doi: 10.1016/S1470-2045(08)70179-7. Epub 2008 Jul 17. PMID 18639491
- [Background] Dutch Comprehensive Cancer Centre. Breast cancer survival in the Netherlands. 2011. Ref Type: Report
- [Background] Basson R, Leiblum S, Brotto L, Derogatis L, Fourcroy J, Fugl-Meyer K, Graziottin A, Heiman JR, Laan E, Meston C, Schover L, van Lankveld J, Schultz WW. Revised definitions of women's sexual dysfunction. J Sex Med. 2004 Jul;1(1):40-8. doi: 10.1111/j.1743-6109.2004.10107.x. PMID 16422982
- [Background] Beckmann J, Johansen L, Richardt C, Blichert-Toft M. Psychological reactions in younger women operated on for breast cancer. Amputation versus resection of the breast with special reference to body-image, sexual identity and sexual function. Dan Med Bull. 1983 Dec;30 Suppl 2:10-3. No abstract available. PMID 6673909
- [Background] Bloom JR, Stewart SL, Chang S, Banks PJ. Then and now: quality of life of young breast cancer survivors. Psychooncology. 2004 Mar;13(3):147-60. doi: 10.1002/pon.794. PMID 15022150
- [Background] Gilbert E, Ussher JM, Perz J. Sexuality after breast cancer: a review. Maturitas. 2010 Aug;66(4):397-407. doi: 10.1016/j.maturitas.2010.03.027. Epub 2010 May 2. PMID 20439140
- [Background] Fobair P, Stewart SL, Chang S, D'Onofrio C, Banks PJ, Bloom JR. Body image and sexual problems in young women with breast cancer. Psychooncology. 2006 Jul;15(7):579-94. doi: 10.1002/pon.991. PMID 16287197
- [Background] Ganz PA, Desmond KA, Belin TR, Meyerowitz BE, Rowland JH. Predictors of sexual health in women after a breast cancer diagnosis. J Clin Oncol. 1999 Aug;17(8):2371-80. doi: 10.1200/JCO.1999.17.8.2371. PMID 10561299
- [Background] Ganz PA, Greendale GA, Petersen L, Kahn B, Bower JE. Breast cancer in younger women: reproductive and late health effects of treatment. J Clin Oncol. 2003 Nov 15;21(22):4184-93. doi: 10.1200/JCO.2003.04.196. PMID 14615446
- [Background] Panjari M, Bell RJ, Davis SR. Sexual function after breast cancer. J Sex Med. 2011 Jan;8(1):294-302. doi: 10.1111/j.1743-6109.2010.02034.x. Epub 2010 Sep 23. PMID 21199377
- [Background] Sadovsky R, Basson R, Krychman M, Morales AM, Schover L, Wang R, Incrocci L. Cancer and sexual problems. J Sex Med. 2010 Jan;7(1 Pt 2):349-73. doi: 10.1111/j.1743-6109.2009.01620.x. PMID 20092444
- [Background] Schover LR. Premature ovarian failure and its consequences: vasomotor symptoms, sexuality, and fertility. J Clin Oncol. 2008 Feb 10;26(5):753-8. doi: 10.1200/JCO.2007.14.1655. PMID 18258983
- [Background] Bredart A, Dolbeault S, Savignoni A, Besancenet C, This P, Giami A, Michaels S, Flahault C, Falcou MC, Asselain B, Copel L. Prevalence and associated factors of sexual problems after early-stage breast cancer treatment: results of a French exploratory survey. Psychooncology. 2011 Aug;20(8):841-50. doi: 10.1002/pon.1789. Epub 2010 Jun 21. PMID 20568085
- [Background] Broeckel JA, Thors CL, Jacobsen PB, Small M, Cox CE. Sexual functioning in long-term breast cancer survivors treated with adjuvant chemotherapy. Breast Cancer Res Treat. 2002 Oct;75(3):241-8. doi: 10.1023/a:1019953027596. PMID 12353813
- [Background] Fobair P, Spiegel D. Concerns about sexuality after breast cancer. Cancer J. 2009 Jan-Feb;15(1):19-26. doi: 10.1097/PPO.0b013e31819587bb. PMID 19197169
- [Background] Kedde, H and Haastrecht, P. Sexual related health of young women with breast cancer. 2008. Utrecht, Rutger Nisso Groep. Ref Type: Report
- [Background] Krychman ML, Pereira L, Carter J, Amsterdam A. Sexual oncology: sexual health issues in women with cancer. Oncology. 2006;71(1-2):18-25. doi: 10.1159/000100521. Epub 2007 Mar 9. PMID 17347586
- [Background] Burwell SR, Case LD, Kaelin C, Avis NE. Sexual problems in younger women after breast cancer surgery. J Clin Oncol. 2006 Jun 20;24(18):2815-21. doi: 10.1200/JCO.2005.04.2499. PMID 16782919
- [Background] Ganz PA, Rowland JH, Desmond K, Meyerowitz BE, Wyatt GE. Life after breast cancer: understanding women's health-related quality of life and sexual functioning. J Clin Oncol. 1998 Feb;16(2):501-14. doi: 10.1200/JCO.1998.16.2.501. PMID 9469334
- [Background] Baucom DH, Porter LS, Kirby JS, Gremore TM, Wiesenthal N, Aldridge W, Fredman SJ, Stanton SE, Scott JL, Halford KW, Keefe FJ. A couple-based intervention for female breast cancer. Psychooncology. 2009 Mar;18(3):276-83. doi: 10.1002/pon.1395. PMID 18702064
- [Background] Dorval M, Guay S, Mondor M, Masse B, Falardeau M, Robidoux A, Deschenes L, Maunsell E. Couples who get closer after breast cancer: frequency and predictors in a prospective investigation. J Clin Oncol. 2005 May 20;23(15):3588-96. doi: 10.1200/JCO.2005.01.628. PMID 15908669
- [Background] Hawkins Y, Ussher J, Gilbert E, Perz J, Sandoval M, Sundquist K. Changes in sexuality and intimacy after the diagnosis and treatment of cancer: the experience of partners in a sexual relationship with a person with cancer. Cancer Nurs. 2009 Jul-Aug;32(4):271-80. doi: 10.1097/NCC.0b013e31819b5a93. PMID 19444088
- [Background] Huyghe E, Sui D, Odensky E, Schover LR. Needs assessment survey to justify establishing a reproductive health clinic at a comprehensive cancer center. J Sex Med. 2009 Jan;6(1):149-63. doi: 10.1111/j.1743-6109.2008.01005.x. Epub 2008 Sep 24. PMID 18823323
- [Derived] Hummel SB, van Lankveld JJ, Oldenburg HS, Hahn DE, Broomans E, Aaronson NK. Internet-based cognitive behavioral therapy for sexual dysfunctions in women treated for breast cancer: design of a multicenter, randomized controlled trial. BMC Cancer. 2015 Apr 28;15:321. doi: 10.1186/s12885-015-1320-z. PMID 25927495